CLINICAL TRIAL: NCT00639067
Title: Breath Test Assay for the Adjunctive Detection of Lung Cancer
Brief Title: Breath Test for Early Detection of Lung Cancer
Status: Completed | Type: Observational
Sponsor: Menssana Research, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: M08-01; 5R44HL070411-05 (NIH)
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Lung Neoplasms
Keywords: Cancer of Lung; Cancer of the Lung; Lung Cancer; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Asymptomatic High Risk Subjects. Smokers aged >=18 undergoing chest CT.
  Breath collected using Breath Collection Apparatus and analyzed for markers of lung cancer.
  Interventions: Device: Breath Collection Apparatus
- 2: Symptomatic High Risk Subjects Without a Tissue Diagnosis. This group will comprise patients who are undergoing medical evaluation for a pulmonary symptom such as chronic unexplained cough or hemoptysis.
  Breath collected using Breath Collection Apparatus and analyzed for markers of lung cancer.
  Interventions: Device: Breath Collection Apparatus
- 3: Symptomatic High Risk Subjects With a Tissue Diagnosis. This group will be found to include a. lung cancer, and b. diseases other than lung cancer e.g. sarcoidosis, COPD or pulmonary infection.
  Breath collected using Breath Collection Apparatus and analyzed for markers of lung cancer.
  Interventions: Device: Breath Collection Apparatus
- 4: Apparently healthy individuals having no signs and symptoms of lung carcinoma.
  Breath collected using Breath Collection Apparatus and analyzed for markers of lung cancer.
  Interventions: Device: Breath Collection Apparatus

INTERVENTIONS:
Device: Breath Collection Apparatus — Breath collected and analyzed for markers of lung cancer.

SUMMARY:
To demonstrate and validate a breath test for detection of early stage lung cancer that could potentially reduce number of deaths.

DETAILED DESCRIPTION:
This is a multicenter study comparing several groups of subjects with and without lung cancer by CT scan, biopsy and the breath test. The breath test will be performed to validate the methodology and the predictive algorithm that were previously developed.

ELIGIBILITY:
Group 1 - Asymptomatic High Risk Subjects

Inclusion criteria

1. Patient is willing and able to cooperate with study and give signed informed consent to participate.
2. Patient has had (or will have) chest imaging with spiral CT within 7 days of breath test.
3. Age at least 18 years.
4. History of at least 10 pack-years of cigarette smoking.
5. Provide written informed consent prior to admission into the study.

Exclusion criteria

1. Previously documented history of cancer of any site.

Group 2 - Symptomatic High Risk Subjects Without a Tissue Diagnosis

Inclusion criteria

1. Patient is willing and able to cooperate with study and give signed informed consent to participate.
2. Patient does not have a tissue diagnosis of pulmonary disease.
3. Patient is undergoing evaluation for an unexplained pulmonary illness which is clinically consistent with lung cancer. This includes patients with unexplained symptoms (e.g. chronic unexplained cough or hemoptysis), unexplained signs (e.g. weight loss, lymphadenopathy) or unexplained investigations (e.g. an abnormal chest x-ray).
4. Actively smoking patients, as well as never smokers and former smokers are eligible for the study so long as a complete smoking consumption history can be recorded.

Exclusion criteria

1. Previously documented history of cancer of any other site.

Group 3 - Symptomatic High Risk Subjects with a Tissue Diagnosis

Inclusion criteria

1. Patient is willing and able to cooperate with study and give signed informed consent to participate.
2. Patient has a tissue diagnosis of a. lung cancer. or b. pulmonary disease other than lung cancer e.g. sarcoidosis, COPD, or pulmonary infection.
3. A diagnosis of lung cancer is defined as cytologic or histologic confirmation of lung cancer by bronchoscopic/thoracoscopic means, sputum cytology, percutaneous fine needle aspiration biopsy. Patients may have either non-small cell lung cancer or small cell lung cancer.
4. Breath VOC collection will be obtained prior to any invasive procedure e.g. thoracotomy, mediastinoscopy or mediastinotomy.
5. Actively smoking patients, as well as never smokers and former smokers are eligible for the study so long as a complete smoking consumption history can be recorded.

Exclusion criteria

1. Previously documented history of cancer of any other site.

Group 4 - Apparently healthy subjects

Inclusion criteria

1. Willingness to follow protocol requirements as evidenced by written, informed consent.
2. Healthy, male or female subjects, ages 18 and older.
3. Subjects who are non smokers having no signs or symptoms of lung carcinoma

Exclusion Criteria

1. Any active ongoing medical problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1. Asymptomatic High Risk Subjects. Smokers aged >=18 undergoing chest CT
  Group 2. Symptomatic High Risk Subjects Without a Tissue Diagnosis. This group will comprise patients who are undergoing medical evaluation for a pulmonary symptom such as chronic unexplained cough or hemoptysis.
  Group 3. Symptomatic High Risk Subjects With a Tissue Diagnosis. This group will be found to include a. lung cancer, and b. diseases other than lung cancer e.g. sarcoidosis, COPD or pulmonary infection.
  Group 4. Apparently healthy individuals having no signs and symptoms of lung carcinoma.
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the breath test as compared to CT and pathology to support primary lung cancer diagnosis. | 30 days after completion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Phillips, MD, FACP, Principal Investigator — Menssana Research, Inc.
Locations (4):
- United States (4):
  - Christiana Hospital, Newark, Delaware
  - MD Anderson Cancer Center, Orlando, Florida
  - New York University Medical Center, New York, New York
  - Swedish Cancer Institute, Seattle, Washington

REFERENCES:
- [Derived] Phillips M, Bauer TL, Pass HI. A volatile biomarker in breath predicts lung cancer and pulmonary nodules. J Breath Res. 2019 Jun 19;13(3):036013. doi: 10.1088/1752-7163/ab21aa. PMID 31085817
- [Derived] Phillips M, Bauer TL, Cataneo RN, Lebauer C, Mundada M, Pass HI, Ramakrishna N, Rom WN, Vallieres E. Blinded Validation of Breath Biomarkers of Lung Cancer, a Potential Ancillary to Chest CT Screening. PLoS One. 2015 Dec 23;10(12):e0142484. doi: 10.1371/journal.pone.0142484. eCollection 2015. PMID 26698306